CLINICAL TRIAL: NCT00883584
Title: A Phase IIa, Proof of Concept Study to Evaluate the Reduction in Inflammatory Biomarkers and Assess Airway Function Following Administration of IMD-1041 in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: IMD-1041 Chronic Obstructive Pulmonary Disease: Proof of Concept (POC) Study
Acronym: COPD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute of Medicinal Molecular Design, Inc. (Industry)
Responsible Party: Covance CRU Ltd. (Sacha Webber-Cross - Project Manager), Covance CRU Ltd.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IMD-10412003-1
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Last update posted 2009-04-23 (Estimated); Status verified 2009-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Proof of Concept; Inflammatory Markers; Lung Function; Chronic Obstructive Pulmonary Disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — IMD-1041

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): IMD-1041
  Interventions: Drug: IMD-1041
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IMD-1041 — Capsule 4 x 100mg BID (30 minutes after breakfast/dinner) 12 weeks
  Arms: 1
Drug: Placebo — Capsule 4 x 100mg BID (30 minutes after breakfast/dinner) 12 weeks
  Arms: 2

SUMMARY:
COPD is a lung disease in which the lung is damaged, making it hard to breathe. In COPD, the airways/tubes that carry air in and out of the lungs are partly obstructed, making it difficult to get air in and out. COPD gets gradually worse over time. At the moment there is no cure for COPD. The best way to slow the disease is to stop smoking. Current medications are used to alleviate shortness of breath and cough, and to treat infections of the lungs that can worsen COPD.

Institute of Medicinal Molecular Design, Inc. (IMMD), a Japanese Drug Discovery Company is developing a compound code named IMD-1041. IMD-1041 is an investigational drug, meaning it is not yet on the market. It is an IKKb inhibitor developed for the treatment of COPD. Unlike most other medications used for COPD currently, IMD-1041 is in capsule form and needs to be taken twice a day. It is also unlike all other drugs in use because it treats the underlying cause of the symptoms.

The purpose of this study is to see if IMD-1041 has the ability to reduce inflammatory derived symptoms and airway remodelling (changes) by looking at certain changes in chemical levels in the blood and sputum (phlegm).

DETAILED DESCRIPTION:
The dose level of IMD 1041 has been selected based on previous clinical trials. The dose to be studied, 400mg, is considered to be efficacious, and is supported by the clinical data in healthy subjects and type 2 diabetic patients.

Single oral doses of 800 mg and multiple oral doses of 400 mg twice daily of IMD-1041 have been shown to be safe and well tolerated by healthy subjects.

Twice daily doses of 200 mg of IMD-1041 have been shown to be safe and well tolerated when given to diabetic patients for 12 weeks.

A placebo (dummy medication) arm has been selected as it is considered the most reliable method to minimise patient and investigator bias and current COPD guidelines suggest the most useful comparison would be with placebo. Exposure placebo will allow a reliable evaluation of IMD 1041, as well as the adverse events caused by the drug compared to those resulting from the COPD natural course.

All patients will be able to remain on the current medications apart from theophylline which is expected to have effects on IKK beta.

The current treatments for COPD do not include a medication of this mechanism of action, who's main aim is to reduce inflammatory and fibrotic changes which cause the symptoms which current standard COPD medications treat.

The study will last for 12-14 weeks, including a 7 day screening period, visit 0 baseline/randomisation visit, visit 1 and visit 3 for all study spec tests, visit 2 and 4/follow up as either a site or telephone contact to check subject compliance and adverse events.

Prior to selection the Investigator will evaluate the eligibility of patients for entry into the trial by reviewing the patients' medical records against the inclusion/exclusion criteria specified in the protocol.

There will be a potential pre-screening visit up to 3 weeks prior to randomisation. This visit will only be applicable for patients who need to stop the medication theophylline which need to be stopped 2 weeks prior to screening. At this visit potential patients will be provided with the information about study activities and requirements. After signing the informed consent form the patient will be asked to stop the medication and return to the study site for screening at least 2 weeks after the visit.

All patients will attend the clinical site for initial screening up to 7 days prior to randomisation. If the patient has not been 'pre-screened' as described above, they will be given information pertaining to study activities and requirements. After signing the informed consent form evaluations will be performed to confirm the patients' eligibility according to the study protocol. The patients' medical history, physical examination, clinical laboratory tests, electrocardiogram (ECG) tracing, blood pressure, pregnancy screening (women of child bearing potential only) will be performed. Blood will be taken for routine clinical laboratory testing.

Following successful screening, patients will return to the site up to seven days (but at least 1 day) after the screening visit for randomisation. There will be a 50:50 chance of the patient being randomised to either IMD 1041 or placebo of whichever they will remain on for the duration of the study. The following will then happen prior to randomisation:

* Patient asked about current health problems, adverse events and any changes to concomitant medications since screening.
* Vitals signs
* Blood will be taken for clinical lab evaluations and biomarker sampling
* Lung functions
* Induced sputum for biomarker sampling
* 2 questionnaires completed Following all of the above evaluations the patient will be randomised and medication dispensed. (A total of 280 tablets will be dispensed, which equates to 4 weeks supply, plus 56 tablets as spares in case of loss or delayed next visit.)

Visit 1 will occur 4 weeks after visit 0 (+/- 2 days). At this visit the following will occur:

* Patient asked about current health problems, adverse events and any changes to concomitant medications since screening.
* vitals signs
* Blood will be taken for clinical lab evaluations, PK analysis and biomarker sampling
* Lung functions
* Induced sputum for biomarker sampling
* Medication will be dispensed. A total of either 4(224) or 8(448) weeks supply will be dispensed depending on whether or not you will attend the clinical site for visit 3.

Visit 2 will occur 4 weeks after visit 1 (+/- 3 days). This visit will be either on site or over the telephone and will be decided by the Principal Investigator on a case-by-case basis. At this visit the following will occur:

* Patient asked about current health problems, adverse events and any changes to concomitant medications since screening.
* Medication dispensed. A total of 4 weeks supply (224 tablets) will be dispensed for patients who attend the site for this visit.

Visit 3 will occur up to 4 weeks after visit 2 (+/- 3 days). At this visit the following will occur:

* Patient asked about current health problems, adverse events and any changes to concomitant medications since screening.
* vitals signs
* Blood will be taken for clinical lab evaluations, PK analysis and biomarker sampling
* Lung functions
* Induced sputum for biomarker sampling
* 2 questionnaires completed
* All medication return and final accountability documented

Visit 4, the follow up visit will be via telephone and will occur 2 weeks after visit 3 (+/- 3 days). The following will occur:

* Patient asked about current health problems, adverse events and any changes to concomitant medications since screening.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant, non-lactating females aged 40 to 80 years of age at the time of the screening visit. (Women of childbearing potential will be allowed to enter the trial only if they are using one medically approved (i.e., mechanical or pharmacological) contraceptive measure. A female is considered to be of childbearing potential unless she has had an hysterectomy, is at least one year post-menopausal, or has undergone tubal ligation. All women of childbearing potential must have a negative pregnancy test at screening visit and week 12 (Visit 3)
* Patients with a clinical diagnosis of COPD, grade 2 or 3 according to the GOLD guidelines 2007 and stable airway obstruction
* Patients with a post salbutamol FEV1 ≥ 30% of the predicted value, < 80% of the predicted value (i.e., 30% ≤ 100 x observed post-salbutamol FEV1/predicted FEV1 <80%) or who is deemed suitable by the Investigator (at either screening or baseline)
* Post-salbutamol FEV1/forced vital capacity (FVC) <70% (i.e,. 100 x post-salbutamol FEV1/FVC <70%)
* Current, or ex-cigarette smokers with a smoking history of at least 10 pack-years
* Patients who have the ability to produce a viable sputum sample (≤ 50% squamous cells)
* Predominant current diagnosis of smoking related COPD
* Patients who were eligible and able to participate in the trial and who consented to do so in writing after the purpose and nature of the investigation had been explained to them

Exclusion Criteria:

* History or current diagnosis of asthma, allergic rhinitis or atopy. N.B. Misdiagnosed asthma or childhood asthma is acceptable, however must be confirmed by the Investigator
* Eosinophil count >600 cells/mm3
* A respiratory tract infection (including the upper respiratory tract) or COPD exacerbation in the 6 weeks prior to the screening visit
* Patients who have been hospitalised for an acute COPD exacerbation in the 12 months or an exacerbation in the last 3 months which was treated with oral steroids prior to the screening visit
* Use of long-term oxygen therapy (≥15 hours/day)
* Clinically significant respiratory conditions defined as: Known active tuberculosis, History of interstitial lung or pulmonary thromboembolic disease, Pulmonary resection during the past 12 months, History of life-threatening COPD, History of bronchiectasis secondary to respiratory diseases other than COPD (e.g., cystic fibrosis, Kartagener's syndrome, etc), Patients who in the Investigator's opinion may need pulmonary rehabilitation or a thoracotomy during the trial
* Clinically significant cardiovascular conditions defined as: Myocardial infarction during the last 6 months, Unstable arrhythmia which required changes in the pharmacological therapy or other intervention during the last 12 months, or newly diagnosed arrhythmia within the previous 3 months, Hospitalisation within the previous 12 months for heart failure functional classes III (marked limitation of activity and only comfortable at rest) and IV (need of complete rest, confinement to bed or chair, discomfort at any physical activity and presence of symptoms at rest) as per the New York Heart Association
* Patients with any other serious or uncontrolled physical or mental dysfunction at the discretion of the Investigator, which could place the patient at higher risk derived from his/her participation in the study, could confound the results of the trial, or is likely to prevent the patient from complying with the requirements of the trial or completing the trial period
* Patients who are not able to perform reproducible spirometry attempts at the screening visit or during the repeat at baseline
* Clinically relevant abnormalities in the results of laboratory, ECG parameters (QTc > 470 milliseconds), or physical examination at the screening evaluation if the abnormality defines a disease state listed as an exclusion criterion, except for those related to COPD
* Patients with a history of drug and/or alcohol abuse that may prevent compliance with trial activities
* Treatment with any IMP within 3 month prior to screening visit
* Changes to any concomitant therapy either for COPD or any other well-controlled illness within 1 month prior to screening visit
* Treatment with a prohibited medication as detailed in Section 5.8

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-05 (Estimated); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
To assess the ability of IMD-1041 to reduce levels of IL-1β, IL-6, TNF-α and GRO-α in blood and/or sputum | 10-12 months

SECONDARY OUTCOMES:
PAI-1 in induced sputum and PAI-1 and t-PA-PAI complex in blood. Levels of CCL5, IL-8, MMP9, TIMP1, MCP-1 and MPO in induced sputum and/or blood | 10-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul Ford, MB, BS, MRCP, PhD, Principal Investigator — King Edward VII Hospital, Windsor, Berkshire, SL4 3DP, UK
Locations (2):
- United Kingdom (2):
  - King Edward VII Hospital (Imperial College, London), Windsor, Berkshire
  - Medicines Evaluation Unit, Wythenshawe Hospital, Manchester